CLINICAL TRIAL: NCT06380101
Title: Prospective, Single Arm IIA Study to Evaluate the Feasibility of a Standardized Nonessential Amino Acid Restriction (NEAAR) Medical Food in Combination With Total Neoadjuvant Therapy (TNT) for Management of Locally Advanced Rectal Cancer (LARC) NEAAR-LARC
Brief Title: Evaluating a Nonessential Amino Acid Restriction (NEAAR) Medical Food With Total Neoadjuvant Therapy for Locally Advanced Rectal Cancer (LARC)
Acronym: NEAAR-LARC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NEAAR-LARC
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nonessential Amino Acid Restriction (NEAAR) Medical Food (Experimental): This is a single arm study in which all subjects will receive NEAAR medical food.
  Interventions: Other: NEAAR Medical Food

INTERVENTIONS:
Other: NEAAR Medical Food — Standardized non-essential amino acid restricted medical food.

SUMMARY:
This clinical study aims to assess feasibility, safety, tolerability, and compliance of a Nonessential Amino Acid Restriction (NEAAR) medical food in adult patients with locally advanced rectal cancer during standard of care short course radiotherapy followed by standard of care chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the rectum
* Clinical stage II (cT3-4, N-) or Stage III (cT any, N+) based on MRI
* Eligible for total mesorectal excision
* No evidence of distant metastasis
* No prior pelvic radiation therapy
* No prior chemotherapy
* Age ≥18 years

Exclusion Criteria:

* Patients unable to undergo MRI
* Other anticancer or experimental therapy
* Body mass index (BMI) <18.5 kg/m2 or >40 kg/m2
* Serious or refractive cachexia or anorexia
* Insulin-dependent diabetes Taking or needs to take any protein or amino acid containing nutritional supplements (e.g., Ensure®) Patients with a condition where high-fat or fatty food is contraindicated History of confirmed food allergy Active wound or skin graft that would require a significant increase in protein requirements for skin integrity and healing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Rate of CTCAE v5.0 non-hematological Grade 3 and higher diarrhea | During standard of care Short-course radiotherapy and total neoadjuvant therapy, up to approximately 1 year

SECONDARY OUTCOMES:
Proportion of clinical complete response 8 weeks post SCRT-TNT with NEAAR medical food defined by the MSK Regression Schema | approximately 8 weeks after SCRT-TNT with NEAAR medical food intervention
Absolute and relative change from baseline of circulating non-essential amino acids | from baseline up to approximately 8 weeks after SCRT-TNT with NEAAR medical food intervention
Proportion of clinical complete response at Week 4 post SCRT with NEAAR medical food | approximately 4 weeks after SCRT with NEAAR medical food intervention
molecular ctDNA response. | approximately 4 weeks after SCRT with NEAAR medical food intervention and 8 weeks post SCRT-TNT with NEAAR medical food intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Richard R Tuli, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States